CLINICAL TRIAL: NCT04629560
Title: Miracle Fruit Powder for the Treatment of Taste Alterations Secondary to Chemotherapy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mt. Sinai Medical Center, Miami (Other)
Responsible Party: Principal Investigator, Mike Cusnir, Medical Director Cancer Center/Chief of Hematology Oncology, Mt. Sinai Medical Center, Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MIRACLE FRUIT
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Taste, Altered; Dysgeusia
MeSH Terms: conditions — Dysgeusia | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned either to the miracle fruit intervention or to supportive measures at first and later participants will cross over to the other intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Miracle Fruit Arm (Experimental): Patient will be randomly assigned, by a computer generated randomization, to receive one miracle fruit tablet of 100 mg 10-15 minutes before lunch and dinner versus supportive measures.
  Interventions: Drug: Miracle Fruit
- Control Arm (supportive measures only) (No Intervention): standard of care supportive measures

INTERVENTIONS:
Drug: Miracle Fruit — one miracle fruit tablet of 100 mg 10-15 minutes before lunch and dinner versus supportive measures. Patients assigned to receive the miracle fruit will receive written instructions regarding the use of the fruit. Patients should put the fruit tablet or powder in the mouth and gently chew/suck to dissolve and cover the tongue with the powder
  Other Names: supportive care
  Arms: Miracle Fruit Arm

SUMMARY:
Purpose and Objective: Compare the incidence of taste alteration in treatment vs. control arms and Compare weight loss in treatment vs. control arms

DETAILED DESCRIPTION:
After patients is explained all potential risks and study guidelines all patients will be given an ICF to sign if they wish to participate. Once the ICF has been signed by patient approximately between 3-5 days will undergo a screening to determine protocol eligibility. If patients qualifies (eligible) for study patients will be randomly assigned either to the miracle fruit intervention or to supportive measures at first and later participants will cross over to the other intervention

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are the following:

  * Patients over 18 years old with a life expectancy of 3 months or more.
  * Patients with an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
  * At enrollment, patients must be able to take oral medications and food reliably without any risk factors for aspiration.
  * Patients that have received at least 1 cycle of chemotherapy and have at least 1 more cycle planned.
  * Patients receiving the following drug-containing chemotherapy regimens: cyclophosphamide, carboplatin, cisplatinum, gemcitibine, methotrexate, doxorubicin, 5-fluorouracil, paclitaxel, docetaxel, vinorelbine, oxaliplatin, irinotecan and etoposide.
  * Patients receiving radiotherapy at the time of chemotherapy are allowed, with the exception of patients receiving radiotherapy for head and neck tumors
  * Patients with the ability to understand and the willingness to sign a written informed consent document written in English and answer all appropriate questionnaires in English or Spanish. (see Appendix 3)
  * Patients with brain metastases are eligible if neurologically stable after appropriate treatment (surgery and/or radiation).

Exclusion Criteria:

* • Patient that have mechanical obstruction of the alimentary tract.

  * Patients who have developed decreased/altered taste sensation for any reason besides chemotherapy
  * Patients with malabsorption or intractable vomiting.
  * Patients who have extensive dental caries
  * Patients who have poor oral hygiene
  * Patients receiving radiotherapy for head and neck tumors.
  * Previous surgery that included ablation or removal of the olfactory component of the taste.
  * Untreatable oral thrush.
  * Women that are pregnant, nursing or of childbearing potential and unwilling to use contraception, as the effects of the miracle fruit on the developing human fetus are unknown.
  * Patients with an ANC < 500/uL .
  * Patients with poorly controlled diabetes mellitus (DM) as determined by their primary physicians will be excluded from the study. All DM patients will be required to check their blood sugar on their usual home glucose meters at least once a day, prior to the ingestion of the miracle fruit. If the patient does not a glucose meter, we will provide the patient with one. Any case of hypoglycemia (blood sugar below 60) should be reported immediately to the treatment physician and the patient should stop the miracle fruit treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-08-18 (Actual); Primary Completion 2011-06-20 (Actual); Study Completion 2011-06-20 (Actual)

PRIMARY OUTCOMES:
Compare the incidence of taste alteration in treatment vs. control arms | 12 months
  Taste alteration will be assessed using questions from the Wickham questionnaire of taste alterations. Patient responses to these questions will be transformed to a 0 to 100 scale.

SECONDARY OUTCOMES:
Compare weight loss in treatment vs. control arms | 12 months
  Weight loss will be determined by comparing baseline (pre-intervention) weight with on-study weight.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Cusnir, MD, Study Chair — Mount Sinai Medical Center of Florida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Griffin AM, Butow PN, Coates AS, Childs AM, Ellis PM, Dunn SM, Tattersall MH. On the receiving end. V: Patient perceptions of the side effects of cancer chemotherapy in 1993. Ann Oncol. 1996 Feb;7(2):189-95. doi: 10.1093/oxfordjournals.annonc.a010548. PMID 8777177
- [Result] Bernhardson BM, Tishelman C, Rutqvist LE. Self-reported taste and smell changes during cancer chemotherapy. Support Care Cancer. 2008 Mar;16(3):275-83. doi: 10.1007/s00520-007-0319-7. Epub 2007 Aug 21. PMID 17710445
- [Result] Marin Caro MM, Laviano A, Pichard C. Impact of nutrition on quality of life during cancer. Curr Opin Clin Nutr Metab Care. 2007 Jul;10(4):480-7. doi: 10.1097/MCO.0b013e3281e2c983. PMID 17563467
- [Result] Wickham RS, Rehwaldt M, Kefer C, Shott S, Abbas K, Glynn-Tucker E, Potter C, Blendowski C. Taste changes experienced by patients receiving chemotherapy. Oncol Nurs Forum. 1999 May;26(4):697-706. PMID 10337648
- [Result] Halyard MY, Jatoi A, Sloan JA, Bearden JD 3rd, Vora SA, Atherton PJ, Perez EA, Soori G, Zalduendo AC, Zhu A, Stella PJ, Loprinzi CL. Does zinc sulfate prevent therapy-induced taste alterations in head and neck cancer patients? Results of phase III double-blind, placebo-controlled trial from the North Central Cancer Treatment Group (N01C4). Int J Radiat Oncol Biol Phys. 2007 Apr 1;67(5):1318-22. doi: 10.1016/j.ijrobp.2006.10.046. PMID 17394940
- [Result] Kurihara K, Beidler LM. Taste-modifying protein from miracle fruit. Science. 1968 Sep 20;161(3847):1241-3. doi: 10.1126/science.161.3847.1241. PMID 5673432
- [Result] Brouwer JN, van der Wel H, Francke A, Henning GJ. Mieraculin, the sweetness-inducing protein from miracle fruit. Nature. 1968 Oct 26;220(5165):373-4. doi: 10.1038/220373a0. No abstract available. PMID 5684879
- [Result] Yamamoto C, Nagai H, Takahashi K, Nakagawa S, Yamaguchi M, Tonoike M, Yamamoto T. Cortical representation of taste-modifying action of miracle fruit in humans. Neuroimage. 2006 Dec;33(4):1145-51. doi: 10.1016/j.neuroimage.2006.08.009. Epub 2006 Oct 3. PMID 17020807
- [Result] Eton DT, Temple LM, Koffler K. Pilot validation of a self-report outcome measure of complementary and alternative medicine. Explore (NY). 2007 Nov-Dec;3(6):592-9. doi: 10.1016/j.explore.2007.08.004. PMID 18005911